CLINICAL TRIAL: NCT07392268
Title: Clinical Utility and Validation of Novel AI-ENDO System in Endoscopic Submucosal Dissection
Brief Title: Validation of AI-ENDO System in Endoscopic Submucosal Dissection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Hon Chi Yip, Assistant Professor, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRE-2025.198
Record Dates: First submitted 2026-01-28; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Superficial Esophageal, Gastric or Colorectal Lesions
Keywords: Al-ENDO SYSTEM; ENDOSCOPIC SUBMUCOSAL DISSECTION; ESD

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-ENDO assisted ESD (Experimental): ESD performed with AI-ENDO assistance
  Interventions: Device: AI-ENDO system; Procedure: Conventional ESD
- Conventional ESD (Active Comparator): ESD performed as in usual clinical practice
  Interventions: Procedure: Conventional ESD

INTERVENTIONS:
Device: AI-ENDO system — During procedure of AI-ENDO assisted ESD, the AI-ENDO system will be connected to the video output system of the main endoscopy processor, so that real-time video data could be fed to the AI-ENDO system for AI analysis. In ESD procedures with AI-ENDO assistance, an auxiliary monitor would be placed side-by-side to the main endoscopy output monitor. This enables endoscopist to simultaneously take reference to the AI interpreted videos.
  Arms: AI-ENDO assisted ESD
Procedure: Conventional ESD — The ESD procedure would be performed in the same manner as in usual clinical practice. In brief, after identification of the target lesion, submucosal injection will be performed to elevate the submucosal layer from the muscularis propria. Mucosal incision followed by submucosal dissection will be performed using dedicated ESD knives. Countertraction method could be utilized based on the endoscopists' personal preference. After successful resection and ensuring adequate haemostasis, the specimen would be retrieved for pathological evaluation.

SUMMARY:
This study is a pilot trial designed to evaluate the feasibility and safety of Al-ENDO assisted ESD in patients with gastrointestinal superficial lesions. Patients with gastrointestinal superficial lesions are scheduled for conventional ESD will be screened for eligibility. The study consists of a few stages:

1. In the first phase, the Al-ENDO system will be tested in the background of the ESD procedure prospectively, but without interfering the endoscopists. The Al-ENDO system would be installed in the Endoscopy Centre in Prince of Wales Hospital. Real-time video analysis would be conducted in the background without interference of the endoscopists' performance. A total of 30 clinical ESD procedures would be analysed, with the goal of achieving good accuracy of the system. The data obtained from this group of patients would also serve as control group for comparison with the subsequent procedures with Al-ENDO support.
2. The second phase of the study would comprise of a the prospective pilot study which Al-ENDO system would be connected to the endoscopy tower with the auxiliary output monitor placing side-by-side with the endoscopy main monitor. The GUI would be displayed in the auxiliary monitor. This phase aims to demonstrate device and patients' safety throughout the procedure, and a total of 10 patients would be recruited, with the target of ensuring smooth dissection procedure without system interruption of failure. In this phase of the study, only expert endoscopist would be involved in performing the procedure.
3. The third phase of the study comprises of a continuation of the initial pilot study with additional of 20 more patients, so that total of 30 procedures would be performed to compare the clinical outcomes with the control group collected previously.

DETAILED DESCRIPTION:
Gastrointestinal (GI) cancer, including stomach, colorectal, and esophageal cancer, is collectively the most common cancer worldwide and the leading cause of cancer-related death globally. The disease imposes a significant burden in Hong Kong, with more than 6,000 new cases diagnosed annually according to local cancer statistics. Despite substantial advances in understanding its pathology, molecular mechanisms, and therapeutic strategies, the survival rate of advanced GI cancer remains suboptimal, with a 5-year survival rate below 60% for most malignancies.

The introduction of government-led initiatives and international cancer policies has expanded early GI cancer screening programs, enabling more patients to be diagnosed at an earlier stage. Early detection allows for less-invasive and more effective treatment options with improved prognosis and increased curative surgical rates.

Complete tumor resection remains the only curative approach for localized GI cancer. Endoscopic submucosal dissection (ESD), a minimally invasive endoscopic technique, has become an established method for early-stage cancers confined to the mucosal layer. ESD enables en-bloc resection of lesions, achieving lower local recurrence rates compared with conventional endoscopic mucosal resection. It has also demonstrated favorable perioperative outcomes, including shorter operative time, lower complication rates, and reduced hospital stay. In countries where screening programs are well implemented, such as Japan, the number of ESD procedures now exceeds radical gastrectomies, making ESD the preferred treatment modality for early gastric cancer. ESD is also used for the treatment of pre-malignant lesions in the GI tract, preventing progression to invasive cancer.

An ESD procedure involves four main phases: (1) marking of the targeted lesion, (2) submucosal injection to create a protective cushion, (3) circumferential incision, and (4) submucosal dissection and removal of the lesion. Although ESD enables complete resection of lesions regardless of size and has a recurrence rate below 1%, it remains technically demanding and carries risks such as bleeding and perforation. In regions where ESD adoption is lower, the learning curve may exceed several hundred cases before proficiency is achieved. Increasing international guidance and training efforts have encouraged a global expansion in the use of ESD as its clinical benefits become more widely recognized.

Safe and precise dissection of cancerous tissue within the complex gastrointestinal environment is critical. Medical safety events in surgical practice contribute significantly to excess hospital stays, costs, and mortality. ESD is technically challenging, requiring endoscopists to maintain clear visualization of the submucosal layer while preserving a stable endoscopic field. Anatomical complexities such as colon flexures, thin colonic walls, mucosal folds, and peristalsis further increase the difficulty of colorectal ESD and raise the risk of incomplete dissection and perforation. Given these challenges, there is a clear need for advanced technologies that enhance surgical precision and safety through intelligent intraoperative guidance.

To improve surgical quality and patient safety, it is essential to develop systems that learn from expert experience and surgical outcomes, providing real-time insights that help prevent operative errors. Identification of the correct dissection plane, submucosal vessels, and cutting landmarks contributes to safe and complete tumor removal.

An AI-ENDO integrated platform has been developed by the investigators to assist endoscopists in enhancing the safety and efficiency of ESD procedures. The system incorporates multiple intelligent functions:

1. Real-time recognition of ESD surgical phases and performance assessment The AI-ENDO platform analyzes surgical workflow to identify the ongoing procedural phase at each moment. The model was trained on high-quality expert ESD videos collected from Prince of Wales Hospital and externally validated using data from several international centers. The system demonstrated high accuracy, precision, and recall, maintaining consistent performance across datasets. The integrated platform operates with real-time computational efficiency.
2. Real-time identification of safe and dangerous zones during ESD The system performs automated segmentation of intraoperative visual fields, identifying anatomic structures such as mucosa, submucosa, muscle layers, and blood vessels. This enables real-time differentiation between safe dissection zones and areas at higher risk for complications. Validation studies using endoscopic surgical videos demonstrated high segmentation accuracy and low latency, with experiments confirming feasibility during live animal trials. AI assistance was associated with shorter procedural time and reduced bleeding events compared with standard procedures of similar complexity.
3. Intelligent dissection trajectory guidance using reinforcement learning Reinforcement learning and imitation learning methods were incorporated to predict optimal dissection trajectories based on expert surgical demonstrations. The system analyzes surgical context in real time to provide decision support and trajectory prediction. Testing on extensive video datasets demonstrated improved accuracy and generalization compared with existing trajectory prediction frameworks.

Through the integration of these functions, the AI-ENDO multifunctional platform aims to support intraoperative decision-making, reduce adverse events, and shorten the learning curve for ESD procedures.

The purpose of this study is to evaluate the clinical utility and efficacy of the AI-ENDO system in endoscopic submucosal dissection for early gastrointestinal neoplasia. Technical success, clinical success, and post-ESD adverse events will be systematically assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patient with superficial esophageal, gastric or colorectal lesions, scheduled for endoscopic submucosal dissection (ESD).
* Age between 18 and 85.

Exclusion Criteria:

* Patient who refused to participate.
* Other cases deemed by the examining physician as unsuitable for safe treatment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Technical success rate | 1 day
  Defined as the rate of procedure with successful en-bloc, without major intra-operative adverse event.
  Unit of measure: % of procedures

SECONDARY OUTCOMES:
Clinical success rate | 30 days
  Defined as the rate of procedure with pathological R0 resection, without major intra-operative and post-operative adverse event.
  Unit of measure: % of procedures
Total procedure time | 1 day
  Time taken from injection to completion of resection. Unit of measure: minutes
Resected lesion size | 1 day
  Size of the resected lesion. Unit of measure: millimeters (mm)
Lesion location | 1 day
  Location of the lesion in the GI tract. Unit of measure: categorical (location)
Lesion histological type | 30 days
  The pathological type of the resected lesion. Unit of measure: categorical (histology)
NASA Task Load Index | 1 day
  Endoscopist's NASA Task Load Index (NASA-TLX) score for the procedure. Score range 0-100, where higher scores means a higher, more demanding perceived workload.
  Unit of measure: score (0-100)
Overall rate of intraprocedural adverse events | 1 day
  Rate of all intra-procedural adverse event. Unit of measure: % of procedures
Rate of intraprocedural adverse events - partial thickness muscle injury | 1 day
  Rate of partial thickness muscle injury without full thickness perforation occurring intra-procedure.
  Unit of measure: % of procedures
Rate of intraprocedural adverse events - full thickness perforation | 1 day
  Rate of full thickness perforation occurring intra-procedure. Unit of measure: % of procedures
Rate of intraprocedural adverse events - haemorrhage | 1 day
  Rate of major bleeding during procedure causing hemodynamic instability, or require blood transfusion, or causing haemoglobin drop > 2 g/dL.
  Unit of measure: % of procedures
Rate of intraprocedural adverse events - Peritonitis | 1 day
  Rate of inflammation of the peritoneum occurring intra-procedure. Unit of measure: % of procedures
Rate of intraprocedural adverse events - others | 1 day
  Rate of any other intra-procedure adverse event. Unit of measure: % of procedures
Overall rate of post-procedural adverse events | 30 days
  Rate of all post-procedural adverse event. Unit of measure: % of patients
Rate of postprocedural adverse events - Electrocoagulation syndrome | 30 days
  Rate of lectrocoagulation syndrome, which is defined as presence of abdominal pain, and fever / leucocytosis after the procedure.
  Unit of measure: % of patients
Rate of post-procedure adverse events - delayed haemorrhage | 30 days
  Rate of significant bleeding with haemoglobin drop > 2 g/dL, or causing hemodynamic instability, or require blood transfusion, or requiring re-intervention by endoscopy / surgery.
  Unit of measure: % of patients
Rate of post-procedure adverse events - delayed perforation | 30 days
  Rate of delayed perforation occurring after completion of procedure. Unit of measure: % of patients
Rate of post-procedure adverse events - others | 30 days
  Rate of any other adverse events after the procedure. Unit of measure: % of patients
AI-system of latency | 1 day
  Time lag in image interpretation by the AI system at ≥25 frames per second. Unit of measure: milliseconds (ms)
AI system accuracy (pixel accuracy) | 1 day
  Mean pixel-wise accuracy of AI interpretation, expressed as percentage of correctly classified pixels.
  Unit of measure: % accuracy
AI system accuracy (Dice similarity coefficient) | 1 day
  Mean spatial overlap between AI-predicted and ground-truth regions (Dice coefficient).
  Unit of measure: Dice score (0-1)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Faculty of Medicine, the Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Schmoll HJ, Van Cutsem E, Stein A, Valentini V, Glimelius B, Haustermans K, Nordlinger B, van de Velde CJ, Balmana J, Regula J, Nagtegaal ID, Beets-Tan RG, Arnold D, Ciardiello F, Hoff P, Kerr D, Kohne CH, Labianca R, Price T, Scheithauer W, Sobrero A, Tabernero J, Aderka D, Barroso S, Bodoky G, Douillard JY, El Ghazaly H, Gallardo J, Garin A, Glynne-Jones R, Jordan K, Meshcheryakov A, Papamichail D, Pfeiffer P, Souglakos I, Turhal S, Cervantes A. ESMO Consensus Guidelines for management of patients with colon and rectal cancer. a personalized approach to clinical decision making. Ann Oncol. 2012 Oct;23(10):2479-2516. doi: 10.1093/annonc/mds236. PMID 23012255
- [Background] Smyth EC, Nilsson M, Grabsch HI, van Grieken NC, Lordick F. Gastric cancer. Lancet. 2020 Aug 29;396(10251):635-648. doi: 10.1016/S0140-6736(20)31288-5. PMID 32861308
- [Background] Nivatvongs S. Surgical management of early colorectal cancer. World J Surg. 2000 Sep;24(9):1052-5. doi: 10.1007/s002680010148. PMID 11036281
- [Background] Hasuike N, Ono H, Boku N, Mizusawa J, Takizawa K, Fukuda H, Oda I, Doyama H, Kaneko K, Hori S, Iishi H, Kurokawa Y, Muto M; Gastrointestinal Endoscopy Group of Japan Clinical Oncology Group (JCOG-GIESG). A non-randomized confirmatory trial of an expanded indication for endoscopic submucosal dissection for intestinal-type gastric cancer (cT1a): the Japan Clinical Oncology Group study (JCOG0607). Gastric Cancer. 2018 Jan;21(1):114-123. doi: 10.1007/s10120-017-0704-y. Epub 2017 Feb 21. PMID 28224238
- [Background] Chiu PW, Teoh AY, To KF, Wong SK, Liu SY, Lam CC, Yung MY, Chan FK, Lau JY, Ng EK. Endoscopic submucosal dissection (ESD) compared with gastrectomy for treatment of early gastric neoplasia: a retrospective cohort study. Surg Endosc. 2012 Dec;26(12):3584-91. doi: 10.1007/s00464-012-2371-8. Epub 2012 Jun 8. PMID 22678176
- [Background] ASGE TECHNOLOGY COMMITTEE; Kantsevoy SV, Adler DG, Conway JD, Diehl DL, Farraye FA, Kwon R, Mamula P, Rodriguez S, Shah RJ, Wong Kee Song LM, Tierney WM. Endoscopic mucosal resection and endoscopic submucosal dissection. Gastrointest Endosc. 2008 Jul;68(1):11-8. doi: 10.1016/j.gie.2008.01.037. No abstract available. PMID 18577472
- [Background] Teoh AY, Chiu PW, Wong SK, Sung JJ, Lau JY, Ng EK. Difficulties and outcomes in starting endoscopic submucosal dissection. Surg Endosc. 2010 May;24(5):1049-54. doi: 10.1007/s00464-009-0724-8. Epub 2009 Nov 13. PMID 19911227
- [Background] Zhang X, Ly EK, Nithyanand S, Modayil RJ, Khodorskiy DO, Neppala S, Bhumi S, DeMaria M, Widmer JL, Friedel DM, Grendell JH, Stavropoulos SN. Learning Curve for Endoscopic Submucosal Dissection With an Untutored, Prevalence-Based Approach in the United States. Clin Gastroenterol Hepatol. 2020 Mar;18(3):580-588.e1. doi: 10.1016/j.cgh.2019.06.008. Epub 2019 Jun 18. PMID 31220645
- [Background] ASGE Standards of Practice Committee; Storm AC, Fishman DS, Buxbaum JL, Coelho-Prabhu N, Al-Haddad MA, Amateau SK, Calderwood AH, DiMaio CJ, Elhanafi SE, Forbes N, Fujii-Lau LL, Jue TL, Kohli DR, Kwon RS, Law JK, Pawa S, Thosani NC, Wani S, Qumseya BJ. American Society for Gastrointestinal Endoscopy guideline on informed consent for GI endoscopic procedures. Gastrointest Endosc. 2022 Feb;95(2):207-215.e2. doi: 10.1016/j.gie.2021.10.022. Epub 2022 Jan 5. PMID 34998575
- [Background] Pimentel-Nunes P, Libanio D, Bastiaansen BAJ, Bhandari P, Bisschops R, Bourke MJ, Esposito G, Lemmers A, Maselli R, Messmann H, Pech O, Pioche M, Vieth M, Weusten BLAM, van Hooft JE, Deprez PH, Dinis-Ribeiro M. Endoscopic submucosal dissection for superficial gastrointestinal lesions: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - Update 2022. Endoscopy. 2022 Jun;54(6):591-622. doi: 10.1055/a-1811-7025. Epub 2022 May 6. PMID 35523224
- [Background] Weingart SN, Iezzoni LI. Looking for medical injuries where the light is bright. JAMA. 2003 Oct 8;290(14):1917-9. doi: 10.1001/jama.290.14.1917. No abstract available. PMID 14532322
- [Background] Cuschieri A. Nature of human error: implications for surgical practice. Ann Surg. 2006 Nov;244(5):642-8. doi: 10.1097/01.sla.0000243601.36582.18. PMID 17060751
- [Background] Chiu PWY, Yip HC, Xia XF, Chan SM, Ng EKW, Lau JYW. How I do it: Flexible 3-D endoscope for endoscopic submucosal dissection. Dig Endosc. 2019 May;31(3):323-328. doi: 10.1111/den.13315. Epub 2019 Mar 21. PMID 30550632
- [Background] Kim ES, Cho KB, Park KS, Lee KI, Jang BK, Chung WJ, Hwang JS. Factors predictive of perforation during endoscopic submucosal dissection for the treatment of colorectal tumors. Endoscopy. 2011 Jul;43(7):573-8. doi: 10.1055/s-0030-1256339. Epub 2011 Mar 29. PMID 21448852
- [Background] Mizushima T, Kato M, Iwanaga I, Sato F, Kubo K, Ehira N, Uebayashi M, Ono S, Nakagawa M, Mabe K, Shimizu Y, Sakamoto N. Technical difficulty according to location, and risk factors for perforation, in endoscopic submucosal dissection of colorectal tumors. Surg Endosc. 2015 Jan;29(1):133-9. doi: 10.1007/s00464-014-3665-9. Epub 2014 Jul 4. PMID 24993172
- [Background] Cao J, Yip HC, Chen Y, Scheppach M, Luo X, Yang H, Cheng MK, Long Y, Jin Y, Chiu PW, Yam Y, Meng HM, Dou Q. Intelligent surgical workflow recognition for endoscopic submucosal dissection with real-time animal study. Nat Commun. 2023 Oct 21;14(1):6676. doi: 10.1038/s41467-023-42451-8. PMID 37865629
- [Background] Scheppach MW, Yip HC, Chen Y, Yang H, Cao J, Chua T, Dou Q, Meng HML, Yam Y, Chiu PW. Feasibility of real-time artificial intelligence-assisted anatomical structure recognition during endoscopic submucosal dissection. Endosc Int Open. 2025 Jun 17;13:a26158008. doi: 10.1055/a-2615-8008. eCollection 2025. PMID 40611836